CLINICAL TRIAL: NCT00417495
Title: Interest of Sentinel Lymph Node Technique in Women With a Multifocal Breast Cancer - IGASSU-0502
Brief Title: Sentinel Lymph Node Technique in Multifocal Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sylvia GIARD, MD, PhD, Centre Oscar Lambret - LILLE (France)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IGASSU 0502
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: adenocarcinoma, breast, multifocal lesions, surgery
MeSH Terms: conditions — Breast Neoplasms; Adenocarcinoma

INTERVENTIONS:
Behavioral: Sentinel Lymph Node Technique

SUMMARY:
The scope of this trial is to assess the Sentinel Lymph Node Technique in Multifocal Breast Cancer

DETAILED DESCRIPTION:
The sentinel lymph node is located preferentially by:

* association of subareolar injection of technecium and blue dye
* or, in case of blue dye allergy, by the subareolar injection of technecium only
* or, in case of no possibility of radioactive isotope subareolar injection , by blue dye injection only This procedures are made the day before the surgery or the day of the surgery
* This procedure is immediately follows by complete axillary dissection during breast surgery
* The anatomopathologic analysis of the 2 samples (sentinel lymph node and axillary dissection) and the histologic confirmation on the removed tumor of the multifocal nature of the breast cancer correspond to the end of the study for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Multifocal invasive breast cancer
* At least 2 focuses (clinically and/or by mammography or ultrasound)
* Proven by pre-surgical histology (on 1 focus at least)
* Age > 18 years old
* Clinically negative axillary lymph nodes
* No treatment before surgery
* Signature of written informed consent

Exclusion Criteria:

* Multifocality proven after surgery
* Non invasive breast cancer
* Inflammatory breast cancer
* Axillary lymph node
* Metastatic disease
* Previous homolateral breast cancer
* Dementia or alterated mental status
* Pregnant or lactating woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
detection rate of sentinel nodes | surgery

SECONDARY OUTCOMES:
number of sentinel nodes removed | surgery
localisation of the sentinel nodes | surgery

CONTACTS AND LOCATIONS:
Overall Officials: GIARD Sylvia, MD, Principal Investigator — Centre Oscar Lambret
Locations (20):
- France (20):
  - Centre Hospitalier Universitaire, Amiens
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Clinique de Flandre, Coudekerque-Branche
  - Centre Georges-Francois LECLERCQ, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CRLC Val d'Aurelle, Montpellier
  - Hôpital Lariboisière, Paris
  - Hopital Tenon, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Gauducheau, Saint-Herblain
  - Centre Hospitalier Sud Léman Valsérine, Saint-Julien-en-Genevois
  - Hôpital Georges PIANTA, Thonon-les-Bains
  - Centre Claudius Regaud, Toulouse
  - Centre Hospitalier, Valenciennes
  - Institut Gustave Roussy, Villejuif